CLINICAL TRIAL: NCT05233111
Title: Prevention of Posttraumatic Stress: A RCT of Modified Brief Prolonged Exposure Therapy (Brief PE) During Inpatient Rehabilitation Post Spinal Cord Injury (SCI)
Brief Title: Brief Prolonged Exposure Therapy Versus Clinical Standard to Reduce Posttraumatic Stress Post Spinal Cord Injury
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 021-339
Record Dates: First submitted 2022-01-14; First posted 2022-02-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries; PTSD; Post-Traumatic Stress Disorder
Keywords: PTSD; SCI; Spinal Cord Injury; Post-Traumatic Stress Disorder
MeSH Terms: conditions — Spinal Cord Injuries; Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Placebo Comparator): Participants in the Treatment as Usual (TAU) group will not receive Prolonged Exposure therapy, but will instead receive the standard clinical treatment received by all persons with spinal cord injury (SCI) at the rehabilitation facility. TAU participants will complete questionnaires/interviews at 1, 3, and 6 months from Baseline.
  Interventions: Behavioral: Treatment as Usual
- Brief Prolonged Exposure (Experimental): Experimental: Brief Prolonged Exposure Participants will receive Brief PE. Subjects in the Brief Prolonged Exposure (BPE) intervention group will additionally receive 3 total therapy sessions, each lasting about 60 minutes spaced about 1-7 days apart. Sessions include education about common reactions to trauma, breathing retraining, identification of self-care tasks and prolonged (repeated) imaginal exposure to trauma memories. Any missed sessions will be made up by scheduling multiple sessions in subsequent weeks. Individuals in the BPE group will complete a screener and then survey questionnaires/ interviews at 1, 3, and 6 months from Baseline.
  Interventions: Behavioral: Brief Prolonged Exposure Therapy

INTERVENTIONS:
Behavioral: Brief Prolonged Exposure Therapy — Brief PE will include 3 therapy sessions, each lasting approximately 60 minutes.
  Arms: Brief Prolonged Exposure
Behavioral: Treatment as Usual — This may include an evaluation by a licensed psychologist and continued follow-up psychotherapy as needed. Treatment as usual participants will have follow-up assessments at 1, 3, and 6 months.
  Arms: Treatment as Usual

SUMMARY:
This study will examine the use brief prolonged exposure (Brief PE) therapy compared to standard clinical care to reduce posttraumatic distress among people who have had a spinal cord injury and are receiving rehabilitation in an inpatient setting.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial examining the efficacy of brief Prolonged Exposure Therapy (Brief PE) delivered in an inpatient rehabilitation setting post-SCI to reduce PTSD symptoms. The overall goal of this project is to test a Brief PE (three 60-minute sessions) to reduce psychological distress after SCI and to mitigate long-term post-SCI distress including PTSD as well as secondary health outcomes (including depression and general anxiety) at 1, 3, and 6 months from baseline. The intervention group (Brief PE) will be compared to standard clinical care with treatment as usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Admitted to the inpatient rehabilitation hospital diagnosed with a SCI following a traumatic event

Exclusion Criteria:

* Patients in police custody
* Not fluent in the English language
* Severe cognitive impairment
* Patients who are acutely suicidal
* Patients with active psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in PSSI-5: PTSD Symptom Scale - Interview for DSM-5 | Baseline, 1 month, 3 months ,6 months
  Change in PTSD symptoms from baseline to 6 months. Total scale ranges from 0-80 points. Higher score indicates greater severity of symptoms.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 | Baseline, 1 month, 3 months ,6 months
  Change in depressed mood from baseline to 6 months. Scored on a 0-27 scale. Higher score indicates greater severity of issues.
Change in Generalized Anxiety Disorder-7 Item | Time Frame: Baseline, 1 month, 3 months, 6 months
  Change in anxiety scored using a 0-21 scale. Higher score indicates greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Powers, PhD, Principal Investigator — Baylor Scott and White Research Institute-Trauma
Locations (1):
- Kirstie A Jones, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No